CLINICAL TRIAL: NCT07235566
Title: A Phase II Clinical Trial Evaluating the Efficacy and Safety of MRG003 in Combination With Pucotenlimab for the Treatment of EGFR-positive Unresectable Locally Advanced or Metastatic ATC/PDTC
Brief Title: MRG003 and Pucotenlimab to Treat Locally Advanced or Metastatic ATC/PDTC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu Wang, Chief of Head and Neck Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIC-TC
Record Dates: First submitted 2025-09-23; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): MRG003 in combination with pucotenlimab
  Interventions: Drug: MRG003 in combination with pucotenlimab

INTERVENTIONS:
Drug: MRG003 in combination with pucotenlimab — After providing full informed consent and signing the informed consent form, eligible subjects will receive MRG003 2.0 mg/kg and pucotenlimab 200 mg. Pucotenlimab will be administered intravenously on the first day of each treatment cycle (infusion time: 60 min ± 15 min; for the first cycle, the infusion time should not be less than 60 minutes). At least 30 minutes after the completion of the pucotenlimab infusion, MRG003 will be administered (infusion time: 60 min ± 15 min; for the first cycle, the infusion time should not be less than 60 minutes). Patients will receive the combination therapy every three weeks until a treatment discontinuation event as defined in the protocol occurs.

SUMMARY:
This study is a single-arm, open-label, multi-cohort, single-center phase II clinical trial designed to observe and evaluate the efficacy and safety of MRG003 (a EGFR-ADC) in combination with pucotenlimab (a PD-1 inhibitor) for the treatment of EGFR-positive unresectable recurrent or metastatic ATC/PDTC. All patients will receive the combination therapy every three weeks until disease progression or other event as defined in the protocol occurs.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, multi-cohort, single-center phase II clinical trial designed to observe and evaluate the efficacy and safety of MRG003 in combination with pucotenlimab for the treatment of EGFR-positive unresectable recurrent or metastatic ATC/PDTC. The trial will establish two cohorts based on the patient's BRAF V600E mutation status: Cohort 1 (BRAF V600E wild-type) or Cohort 2 (BRAF V600E mutant type). Each cohort will enroll approximately 30 evaluable subjects. After providing full informed consent and signing the informed consent form, eligible subjects will receive MRG003 2.0 mg/kg and Pucotenlimab 200 mg. Patients will receive the combination therapy every three weeks until a treatment discontinuation event as defined in the protocol occurs.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form and comply with the protocol requirements.
* Age ≥18 years on the day of signing the informed consent form, regardless of gender.
* Expected survival time ≥12 weeks.
* Patients with pathologically confirmed EGFR-positive ATC or PDTC, currently in a recurrent or metastatic stage and not eligible for curative resection. ATC/PDTC may coexist with differentiated thyroid cancer. EGFR positivity is defined as >10% of tumor cells showing positive immunohistochemical staining.
* For subjects with either BRAF V600E wild-type or mutant-type, treatment-naive patients or those who have previously received targeted therapy ± immunotherapy are eligible for enrollment. Regarding neoadjuvant/adjuvant therapy, if recurrence occurs within 6 months after completing neoadjuvant/adjuvant therapy, such treatment will be considered as systemic therapy for the recurrent/metastatic stage.
* Subjects must be able to provide tumor tissue specimens (paraffin blocks, paraffin-embedded sections, or fresh tissue sections) from primary or metastatic sites for pathological testing. The most recent archived tumor tissue specimen should be used. If archived tissue is unavailable, a new biopsy must be performed.
* There must be radiographic evidence of disease progression during or after the most recent treatment, confirmed by the investigator. According to RECIST 1.1 criteria, there must be at least one measurable extracranial lesion at baseline. Measurable lesions should not have been irradiated, unless the lesion within a prior radiation field or after local treatment has demonstrated progression.
* Adverse events related to prior anti-tumor treatment have recovered to ≤ Grade 1 according to NCI CTCAE v5.0 (except for alopecia, non-clinically significant or asymptomatic laboratory abnormalities).
* ECOG performance status of 0 or 1 within 7 days prior to treatment.
* No severe cardiac dysfunction, with left ventricular ejection fraction (LVEF) ≥50% within 28 days prior to treatment.
* Organ function levels must meet the following requirements within 7 days prior to treatment.
* Fertile male and female subjects of childbearing potential must agree to use effective contraception from the time of signing the informed consent form until 6 months after the last dose of the study drug. Women of childbearing potential include premenopausal women and women within 2 years of menopause. A negative serum pregnancy test result within ≤7 days prior to the first dose of the study drug is required for women of childbearing potential.

Exclusion Criteria:

* Medullary thyroid carcinoma or other malignancies not originating from thyroid follicular cells;
* History of other primary malignancies; Except for basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix; or patients who have received radical treatment and have had no recurrence within 5 years may participate in this trial;
* Received any of the following treatments:

  1. Prior treatment with an ADC drug;
  2. Treatment with an investigational drug from another clinical trial within 28 days prior to the first dose (excluding already marketed drugs);
  3. Treatment with anti-tumor Chinese patent medicines or herbal medicines within 14 days prior to the first dose;
  4. Radiotherapy within 28 days prior to the first dose, or palliative radiotherapy for bone metastases within 2 weeks prior to the first dose;
  5. Major surgery within 28 days prior to the first dose without full recovery, or planned major surgery within the first 12 weeks after receiving the study drug.
* Untreated or unstable brain parenchymal metastases, spinal cord metastases or compression, carcinomatous meningitis, or leptomeningeal metastases; Note: Patients who have received local brain therapy may be enrolled if brain imaging shows stability for at least 28 days prior to the first dose, with no evidence of cerebral edema and no requirement for corticosteroid therapy.
* Presence of third-space fluid that cannot be controlled by methods such as drainage (e.g., massive ascites, pleural effusion, pericardial effusion, etc.), or subjects who required drainage to control third-space fluid within 14 days prior to dosing;
* Any severe or uncontrolled systemic disease, in the investigator's judgment, including poorly controlled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg), poorly controlled diabetes, signs of active bleeding, etc.;
* Poorly controlled cardiac disease, including heart failure of NYHA class II or above, unstable angina, myocardial infarction within the past year, clinically significant supraventricular or ventricular arrhythmia requiring treatment, or long QT syndrome, such as QTcF > 450 ms (men) or QTcF > 470 ms (women);
* Evidence of active infection, including hepatitis B (requiring both HBsAg positivity and HBV DNA ≥2000 IU/ml, excluding hepatitis due to drugs or other causes), hepatitis C (requiring both anti-HCV antibody positivity and HCV RNA above the lower limit of detection), or human immunodeficiency virus (HIV) infection; uncontrolled active bacterial, other viral, fungal, rickettsial, or parasitic infections, unless treated and resolved prior to study drug administration;
* History of allergy to any component of pucotenlimab or MRG003 (histidine, histidine hydrochloride, sucrose, mannitol, and polysorbate 80), or history of ≥ Grade 3 allergy to macromolecular protein preparations/monoclonal antibodies;
* History of primary immunodeficiency or active autoimmune disease, currently using immunosuppressants or systemic hormonal therapy (at a dose ≥10 mg/day of prednisone or equivalent), and continuing use within 2 weeks prior to enrollment;
* Positive serum pregnancy test or lactating women who are unwilling to use adequate contraception during the study and for 6 months after the end of study drug treatment;
* Any other situation considered by the investigator as unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate，ORR | 2 years
  Objective Response Rate (ORR) as assessed based on RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China